CLINICAL TRIAL: NCT06304025
Title: Pilot Study: Sequential Administration of Allogeneic Mesenchymal Stem Cells Thawed or Expanded in Vitro for the Treatment of Acute Graft-versus-host Disease Refractory to Second Line Treatment
Brief Title: Sequential Administration of WJ-MSCs for the Treatment of GvHD Refractory to Second Line Treatment
Acronym: GvHD
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle (Other)
Collaborators: Instituto Distrital de Ciencia, Biotecnología e Innovación en Salud - IDCBIS (Other)
Responsible Party: Principal Investigator, Martha Ligia Arango Rodríguez, Scientific technical director of the Center for advanced therapies Fundación Oftalmológica de Santander (FOSCAL), Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GvHD 01
Record Dates: First submitted 2024-01-19; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Graft Versus Host Disease
Keywords: Graft-versus-host Disease; Ruxolitinib; Mesenchymal Stem Cells
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Intervention Model Description: Experimental (pilot clinical study), randomized, blind, and parallel.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thawed allogeneic WJ-MSCs (Experimental): Administration intravenously of 1x106 cells/kg weight of thawed allogeneic WJ-MSCs
  Interventions: Biological: Wharton's jelly mesenchymal stem cells (WJ-MSCs)
- Expanding allogeneic WJ-MSCs (Experimental): Administration intravenously of 1x106 cells/kg weight of expanding allogeneic WJ-MSCs
  Interventions: Biological: Wharton's jelly mesenchymal stem cells (WJ-MSCs)

INTERVENTIONS:
Biological: Wharton's jelly mesenchymal stem cells (WJ-MSCs) — Four doses of 1x10 6 of thawed allogeneic WJ-MSCs or expanding allogeneic WJ-MSCs / kg at 1, 4, 11, and 18 days

SUMMARY:
Hematopoietic stem cell transplantation (HSCT) is the treatment of choice for malignant hemopathies, but highlights the limitations of long-term results due to the high toxicity of the procedure and the development of Graft versus Host Disease (GVHD). Conventional treatments for GVHD have limited success rates, and some patients may be refractory to ruxolitinib, a second-line treatment option. As a result, there is a need to explore alternative immuno-modulatory therapies, such as the use of Wharton's jelly mesenchymal stem cells (WJ-MSCs).

The research question aims to investigate the safety and potential benefits of sequentially infusing thawed or expanding allogeneic WJ-MSCs in the treatment of acute GVHD refractory to second-line treatment in patients from the Colombian population. This pilot clinical study is being conducted to address the unmet need for patients who develop GVHD resistant to ruxolitinib.

DETAILED DESCRIPTION:
In recent decades, the number of HSCTs has significantly increased, as it is considered the ideal therapeutic approach for a wide range of hematological diseases. However, GVHD is the most common and severe complication following transplantation, and it remains the major limiting factor for the success of HSCT. It has been reported that the incidence of acute GVHD is approximately 50% in patients who receive HSCT from an HLA-matched donor, and it increases in cases of HLA-mismatched donors, despite having prophylactic treatment. Patients who develop GVHD have a poor prognosis, with a survival rate ranging from 5-25% depending on the severity of the disease. This is strongly related to the lack of effective treatments. In addition to the high morbidity and mortality, GVHD represents a significant financial burden for public healthcare systems worldwide. A recent study in 2018 in the United States reported that the cost of complete remission for a 6-month period with ruxolitinib, one of the most commonly used treatments for both acute and chronic GVHD, was $1,187,657 USD.

In this context, the American Society for Blood and Marrow Transplantation considers MSCs as a prominent therapeutic tool for the treatment of GVHD, as they significantly improve both the symptoms of the most frequently affected organs (skin, liver, and intestines) and the treatment response parameters and overall survival. Colombia is not exempt from this issue; the rise of HSCT in our country is evident. Therefore, the development of a novel and effective therapeutic strategy for GVHD is a priority and demands further scientific research.

Finally, with the development of this pilot study, the aim is to lay the groundwork for conducting medium- and large-scale clinical trials in our Colombian population, where clinical studies with this type of therapeutic approach have not yet been conducted.

ELIGIBILITY:
Inclusion criteria:

* Aged between 18 and 65 years.
* With a diagnosis of malignant hemopathies, who have undergone allogeneic HSCT and who are diagnosed with acute GVHD refractory to second-line treatment.
* Patients who have received bone marrow and/or peripheral blood as a source of cells.
* Patients who have received cells from a family or unrelated donor
* Myeloablative or non-myeloablative conditioning method.
* Adequate cardiac function without evidence of uncontrolled hypertension, congestive heart failure, angor pectoris, or acute myocardial infarction in the 6 months prior to the process.
* Adequate lung function without evidence of severe obstructive or restrictive lung disease.
* Informed consent signed by the patient.

Exclusion Criteria:

* Patients from the Transplant Unit of the FOSCAL.
* Patients with a diagnosis of hemopathy that has not been controlled by the transplant or is progressing at the time of treatment.
* Bacterial, viral, or fungal infection that is not being controlled with adequate treatment.
* Cardiac and/or pulmonary function in uncontrolled altered conditions.
* According to medical criteria, patients who are not in an adequate situation to tolerate the treatment.
* Pregnant women or women at risk of pregnancy due to inadequate contraceptive measures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events: safety and tolerability | 12 months
  The trial's primary endpoint is to determine the safety of WJ-MSCs administration; for that, we will assess the number of treatment-related adverse events (AEs) reported according to the Common Terminology Criteria for AE classification and presentation of infectious complications after administration of WJ-MSCs.
Efficacy clinic profile: response of acute GVDH | 12 months
  • Response of acute GVHD refractory to second-line treatment (yes or no).
Efficacy clinic profile : duration of response | 12 months
  • Duration of response/incidence of relapses( time: days or months).
Efficacy clinic profile: decrease in treatments | 12 months
  • Decrease in corticosteroids or concomitant immunosuppressive treatment (dose).
Efficacy biological profile: secretion pattern of soluble factors | 12 months
  • Evolution of the secretion pattern of the following soluble factors: cytokines CK8, Reg3α, Elafina, ST2, INF-γ, TNF-α, IL-12, IL-10, CXCL-9 and CXCL-10 (concentration: mg or μg or pg or others).
Efficacy biological profile: cell populations | 12 months
  • Determination of the following cell populations: T lymphocytes, Naive, B lymphocytes, dendritic cells, and Natural Killer cells in blood pre and post-treatment with WJ-MSCs (percentage).
Efficacy biological profile: ocrrelation of the biological markers with the clinical response | 12 months
  • Correlation of the profile of biological markers with the clinical response (-1 and 1).

IPD SHARING:
Plan to Share IPD: No